## Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD)

#### Informed Consent Form Version 7.2 dated 17NOV2021

#### **Principal Investigators:**

Kimford J. Meador, M.D. Stanford University Palo Alto, California

Page B. Pennell, M.D.
Harvard Brigham & Women's Hospital
Boston, Massachusetts

Data and Statistical Center PI: Abigail Matthews, Ph.D. The Emmes Corporation Rockville, Maryland

#### Supported by:

The National Institute of Neurological
Disorders and Stroke (NINDS) & Eunice Kennedy Shriver National Institute of Child
Health and Human Development (NICHD)

Grant #1U01-NS038455

NCT 01730170

IRB Use Only
Approval Date: November 30, 2022
Expiration Date: November 30, 2023

Protocol Director: Kimford Meador, MD

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

| Please check all that are applicable: |
|------------------------------------------|
| $\ \ $ |
| Print your name here: |
| $\ \ $ |
| Print child's name here: |

#### FOR QUESTIONS ABOUT THE STUDY, CONTACT:

Department of Neurology & Neurological Sciences Stanford Comprehensive Epilepsy Center Stanford University School of Medicine 213 Ouarry Road

Dr. Kimford Meador

Palo Alto, California 94304

(650) 725-6648

**DESCRIPTION:** You are being asked to continue participating in a research study. This form is designed to tell you everything you need to think about before you decide to consent (agree) continue in the study or not to be in the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. You can skip any questions that you do not wish to answer.

Our preliminary genetic analyses are providing interesting findings, but we are concerned that we will run out of genetic samples before completing all of our future genetic studies. We are requesting to collect an additional genetic sample from you and your child.

Before making your decision:

- Please carefully read this form or have it read to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. By signing this form you will not give up any legal rights.

IRB Use Only
Approval Date: November 30, 2022
Expiration Date: November 30, 2023

Protocol Director: Kimford Meador, MD

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You may search this Web site at any time.

**STUDY OVERVIEW:** Mothers with epilepsy, mothers without epilepsy, and their children are being asked to continue in this project. You are being asked to participate in this project because you are currently enrolled or have been enrolled in the MONEAD study. You cannot participate in a clinical trial at the same time you participate in this study. You will be one of approximately 451 women and their children to continue in this study in the study at 20 clinical sites across the United States.

Yours or your child's medical care and treatment will not be altered in any way for this study. Your participation in this study will not change your treating obstetrician, neurologist, primary care physician, or pediatrician. You will receive no medications or other types of treatment as part of this study. You will be asked to agree to have medical records such as your medical history, obstetrical, delivery, and pediatric records released to the study staff.

**PROCEDURES:** You and your child's participation will require up to 4 visits and 16 telephone contacts depending on how old your child is currently. Occasionally, your interview with a research assistant might be audio/videotaped so that we can make sure our research assistants are scoring these standard scales the same way each time. These interviews will be labeled with a study number, stored in a locked cabinet and destroyed at the conclusion of the study.

When your child is 15, 18 & 21 months, you will be contacted by the study staff by telephone. You will not have to come into the study offices, but completing the telephone interviews are just as important to the study. During these calls, you will be asked if you and your child had any health problems and if you are continuing, changing, or starting new medications since the last visit.

When your child is 24 months (2 years) of age (Visit 9), you will be asked if you and your child had any health problems. You will be asked to complete questionnaires on changes in employment, your stress levels, and mood, and your child's development. You will be asked to complete questionnaires about your child's behavior. Your child will have a physical and neurological exam and have a test of behavior and thinking abilities. Your child's handedness will be evaluated. If the assessments show any cause for concern, your child will be referred for further testing and follow-up.

When your child is 27, 30, and 33 months of age you will be contacted by the study staff by telephone. You will not have to come into the study offices, but completing the telephone interviews are just as important to the study. During these calls, you will be asked if you and your child had any health problems.

When your child is 36 months (3 years) of age (Visit 10) you will be asked if you and your child had any health problems. You will be asked to complete questionnaires on your stress

IRB Use Only
Approval Date: November 30, 2022
Expiration Date: November 30, 2023

Protocol Director: Kimford Meador, MD

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

levels and mood, your child's development. You will be asked to complete questionnaires about your child's behavior. Your child will have a physical and neurological exam and have tests of behavior and thinking abilities. Your child will also have testing of memory, logic, and motor skills performed. Your child's handedness will be evaluated. The assessments should not take more than 2 hours. If the assessments show any cause for concern, your child will be referred for counseling and follow-up.

When your child is 39, 42, 45, 48, and 51 months of age you will be contacted by the study staff by telephone. You will not have to come into the study offices, but completing the telephone interviews are just as important to the study. During these calls, you will be asked if you and your child had any health problems.

When your child is 54 months (4  $\frac{1}{2}$  years) of age (Visit 11) you will be asked if you and your child had any health problems. You will be asked to complete questionnaires on your stress levels and mood, your child's development. You will be asked to complete questionnaires about your child's behavior. Your child will have a physical and neurological exam and have a test of creative thinking. This assessment should not take more than an hour.

When your child is 57, 60, 63, 66, and 69 months of age you will be contacted by the study staff by telephone. You will not have to come into the study offices, but completing the telephone interviews is just as important to the study. During these calls, you will be asked if you and your child had any health problems.

When your child is 72 months (6 years) of age (Visit 12) you will be asked if you and your child had any health problems. You will be asked to complete questionnaires on your stress levels and mood, your child's development. You will be asked to complete questionnaires about your child's behavior. Your child will have a physical and neurological exam and have tests of behavior and thinking abilities. Your child will also have testing of memory, logic, and motor skills performed. Your child's handedness will be evaluated. The assessments should not take more than 6 hours. This testing session will include a break for your child and, if necessary, can be split over 2 days. If the assessments show any cause for concern, your child will be referred for counseling and follow-up.

Occasionally, your interview with a research assistant might be audio/videotaped so that we can make sure our research assistants are scoring these standard scales the same way each time.

| I give consent to | be aud | lio/videotaped | during | this study |
|-------------------|--------|----------------|--------|------------|
| Please initial: | Yes | No | | |

If you provide permission, your child's teacher will be asked to participate in the study as well. The teacher's involvement will consist of filling out a questionnaire about your child's behavior.

It is important that you report any hospitalizations, illnesses or other health problems you may have to the study staff at any time while you are participating in the study. If you are taking

IRB Use Only

Approval Date: November 30, 2022 Expiration Date: November 30, 2023

Protocol Director: Kimford Meador, MD

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

medications, you may be asked to bring a container of each in so the study staff may obtain accurate information about its dose and how often you should take it.

You have previously provided the project a genetic sample by blood draw, heel stick or swabbing. The goal is to increase the amount of sample we have already collected to ensure there is enough for possible future research projects investigating any enzymes or genetic susceptibility in the subjects that interact/work with AED metabolism and if those are related to any mother or child outcomes.

You will rub a cotton swab firmly against the inside of your and your child's cheek to collect this sample. Each will use a separate swab. If you are not comfortable doing this yourself, the study staff can do the collection for you.

We plan to perform genetic research using you and your child's tissue samples that have been collected. All living things are made of cells. DNA is the material in cells that makes up your genes which contain the instructions telling our bodies how to grow, work, and determine physical characteristics such as hair and eye color. Genes are passed from parent to child. As we do not yet know which genes fit our current hypotheses about how anti-epileptic medications may impact early development in exposed infants, we will utilize continually improving DNA sequencing technologies for our studies. Your genetic information may be shared with other investigators in other study groups. The swab samples will be stored at the University of Minnesota. The genetic data will be coded to protect your identity.

Check ONE answer below:

Even if you initially agree to participate, later you can have your sample destroyed if you change your mind and decide you do not want to participate by notifying your study doctor in writing.

| Yes, studies. | I agree to participate and to allow my child to participate in the project's genetic |
|---|---|
| Yes, | I agree to participate but I do not want my child to participate. |
| Yes, | I agree to allow my child to participate, but I do not want to participate. |
| No, I project. | I do not want myself or my child to participate in the genetic sampling in this |

If you are coming in-person to research visits, you are required to be fully vaccinated—2 doses (1 for Johnson and Johnson), 2 weeks out and to provide proof of your vaccination (e.g., CDC COVID-19 Vaccination Card, e-Health record, etc.) to the researcher prior to study participation. Alternately, you can provide a negative COVID test within 72 hours of your visit.

IRB Use Only
Approval Date: November 30, 2022
Expiration Date: November 30, 2023

Protocol Director: Kimford Meador, MD

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

**RISKS AND BENEFITS:** The main risks of participation are fatigue and feelings of unease answering questions. Your child may become restless with the tests and questions. We will make every attempt to schedule and perform the tasks so as to reduce these risks. You and your child may refuse to answer any question that upsets you. Side effects and problems not listed above and not expected at this time may occur. You will be told of any changes in the way the study is done and of any risks to you or your child.

This study is not designed to benefit you directly. The study results may be used to help others in the future. We cannot and do not guarantee or promise that you will receive any benefits from this study. It is possible that the researchers will learn something new during the study about the risks of being in it. If this happens, they will tell you about it. Then you can decide if you want to continue to be in this study or not. You may be asked to sign a new consent form that includes the new information if you decide to stay in the study.

Your decision whether or not to participate in this study will not affect your employment/medical care.

You and/or your child may feel some discomfort when taking the samples.

**Confidentiality:** The Data Management Center located at The EMMES Corporation in Rockville, Maryland is the company that developed and maintains the electronic database where information collected in the study is entered and stored for analysis. Although no information that identifies you is entered into this database, The EMMES Corporation will send out representatives to each center in the study to review the information collected and to make sure that the data is being collected and entered correctly. A study number rather than your name will be used on study records wherever possible. Your name and other facts that might point to you will not appear when we present this study or publish its results.

**TIME INVOLVEMENT:** Your participation, and that of your child, in this experiment will take approximately 4 years.

**PAYMENTS:** You will be paid for each completed study visit as noted in the following table:

| Visit/Telephone Contact | Stipend |
|----------------------------------------------------------|--------------|
| Visits 8a, 8b, 8c (15, 18, & 21 mo.) | \$15 each 45 |
| Visit 9 (2 yr.) | \$200 |
| Visits 9a, 9b, 9c (27, 30, & 33 mo.) | \$15 each 45 |
| Visit 10 (3 yr.) | \$300 |
| Visits 10a, 10b, 10c, 10d, 10e (39, 42, 45, 48 & 51 mo.) | \$15 each |
| Visit 11 (4 ½ yr.) | \$300 |
| Visit 11a, 11b, 11c, 11d, 11e (57, 60, 63, 66, & 69 mo.) | \$15 each |
| Visit 12 (6 yr.) | \$500 |

IRB Use Only

Approval Date: November 30, 2022 Expiration Date: November 30, 2023

Protocol Director: Kimford Meador, MD

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

If you do not finish the study, you will not be paid for the visits you have not completed. You will receive \$1,540 total, if you complete all study visits.

We will also give your child an age appropriate card or toy at their 2, 3, 4 ½ and 6 YO visits.

Periodically you will receive a study related newsletter.

You will receive a stipend of \$15 for each sample collected from the you and your child(ren).

Payments may only be made to U.S. citizens, legal resident aliens, and those who have a work eligible visa. You may need to provide your social security number to receive payment.

**PARTICIPANT'S RIGHTS:** If you have read this form and have decided to participate in this project, please understand your participation is voluntary and you have the right to withdraw your consent or discontinue participation at any time without penalty or loss of benefits to which you are otherwise entitled.

The results of this research study may be presented at scientific or professional meetings or published in scientific journals. However, your identity will not be disclosed. You have the right to refuse to answer particular questions.

IRB Use Only Approval Date: November 30, 2022 Expiration Date: November 30,

Kimford Meador, MD Protocol Director:

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

## Authorization To Use Your Health Information For **Research Purposes**

Because information about you and your health is personal and private, it generally cannot be used in this research study without your written authorization. If you sign this form, it will provide that authorization. The form is intended to inform you about how your health information will be used or disclosed in the study. Your information will only be used in accordance with this authorization form and the informed consent form and as required or allowed by law. Please read it carefully before signing it.

## What is the purpose of this research study and how will my health information be utilized in the study?

Most Women with epilepsy have normal pregnancies, but appear to be at risk for problems during pregnancy (e.g., seizures, change in medications, depression, csections) and adverse outcomes in their children (e.g., thinking or behavioral problems). The purpose of this observational study is to establish the risk and determine the factors or contributions to those risks.

If you sign this form, you give us your permission to use your PHI for the conduct and oversight of this research study. Your health information may be used in future publications.

## Do I have to sign this authorization form?

You do not have to sign this authorization form. But if you do not, you will not be able to participate in this research study.

Signing the form is not a condition for receiving any medical care outside the study.

## If I sign, can I revoke it or withdraw from the research later?

If you decide to participate, you are free to withdraw your authorization regarding the use and disclosure of your health information (and to discontinue any other participation in the study) at any time. After any revocation, your health information will no longer be used or disclosed in the study, except to the extent that the law allows us to continue using your information (e.g., necessary to maintain integrity of research). If you wish to revoke your authorization for the research use or disclosure of your health information in this study, you must write to: Dr. Kimford Meador at 213 Ouarry Road, Palo Alto CA 94304.

Approval Date: November 30, 2022 Expiration Date: November 30, 2023

IRB Use Only

Protocol Director: Kimford Meador. MD

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

## What Personal Information Will Be Obtained, Used or Disclosed?

Your health information related to this study, may be used or disclosed in connection with this research study, including, but not limited to, your medical and psychiatric history; HIV or VDRL status, demographics such as age, educational achievements, employment status and physical factors such as height, weight, measurement of the size of your head, and imaging results. Other PHI may include your mental health status, alcohol, drug and tobacco use. Information about your child's delivery, health and development will be used. You and your child's medical records from your primary care physician, neurologist, obstetrician and pediatrician will be used to collect or confirm this information. Upon agreement, your voice may be recorded on videotape to evaluate the study assessor's performance submitted to the Psychiatry Core. Other PHI to be collected may include outside assessments/diagnoses of autism and/or developmental delay, child interventions such as Early Intervention, Head Start and Special Education services and information about your mental health status.

### Who May Use or Disclose the Information?

The following parties are authorized to use and/or disclose your health information in connection with this research study:

- The Protocol Director Dr. Kimford Meador
- The Stanford University Administrative Panel on Human Subjects in Medical Research and any other unit of Stanford University as necessary
- Research Staff

## Who May Receive or Use the Information?

The parties listed in the preceding paragraph may disclose your health information to the following persons and organizations for their use in connection with this research study:

- The Office for Human Research Protections in the U.S. Department of Health and Human Services
- The study's funding institution, Emory University
- National Institute of Neurological Disorders and Stroke/Eunice Kennedy Shriver National Institute of Child Health and Human Development are the Sponsors of this Research. The Sponsor(s) may use and disclose your PHI to make sure the research is done correctly. They may also use your PHI to collect and analyze the results of the research. The Sponsor may have other

IRB Use Only
Approval Date: November 30, 2022
Expiration Date: November 30, 2023

Protocol Director: Kimford Meador, MD

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

people and groups help conduct, oversee, and analyze the study. These people or groups will use your PHI.

- The following groups may also use and disclose your PHI. They will do this to make sure the research is done correctly and safely. The groups are:
  - o the Emory University Institutional Review Board
  - o the Emory University Office of Research Compliance
  - research monitors and reviewers
  - The EMMES Corporation, the Data & Statistical Center.
  - the Office for Human Subjects Research Protections the FDA, and the National Institutes of Health
  - o public health agencies
  - University of Arkansas, Psychiatry Core

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

Your information may be re-disclosed by the recipients described above, if they are not required by law to protect the privacy of the information.

## When will my authorization expire?

Your authorization for the use and/or disclosure of your health information will end on January 1, 2050 or when the research project ends, whichever is earlier.

# Description of Representative's Authority to Act for Subject Will access to my medical record be limited during the study?

To maintain the integrity of this research study, you may not have access to any health information developed as part of this study until it is completed. At that

IRB Use Only

Approval Date: November 30, 2022 Expiration Date: November 30, 2023

Protocol Director: Kimford Meador, MD

(e.g., parent, guardian or conservator)

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

point, you would have access to such health information if it was used to make a

medical or billing decision about you (e.g., if included in your official medical record).

Signature of Adult Participant

Date

Print Name of Adult Participant

Signature of Legally Authorized Representative (LAR)

(e.g., parent, guardian or conservator)

Print Name of LAR

LAR's Authority to Act for Participant

IRB Use Only Approval Date: November 30, 2022

Expiration Date: November 30,

Protocol Director: Kimford Meador, MD

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

#### WITHDRAWAL FROM STUDY

You have the right to leave a study at any time without penalty. You may refuse to do any procedures you do not feel comfortable with, or answer any questions that you do not wish to answer.

The Protocol Director may also withdraw you from the study without your consent for one or more of the following reasons:

- Failure to follow the instructions of the Protocol Director and study staff.
- The Protocol Director decides that continuing your participation could be harmful to you.
- You were to object to any future changes that may be made in the study plan
- The study is cancelled.
- Other administrative reasons.
- Unanticipated circumstances.

You have the right to refuse to allow the investigators to share your sample at any time without penalty. If you change your mind, you may be able to withdraw the remaining sample at a later time by notifying the MONEAD staff.

#### **CONTACT INFORMATION:**

If you have any questions, concerns or complaints about this research study, its procedures, risks and benefits, or alternative courses of treatment, you should ask the Protocol Director, Dr. Kimford Meador, at (650) 725-6648. You should also contact him at any time if you feel you have been hurt by being a part of this study.

Independent Contact: If you are not satisfied with how this study is being conducted, or if you have any concerns, complaints, or general questions about the research or your rights as a participant, please contact the Stanford Institutional Review Board (IRB) to speak to someone independent of the research team at (650) 723-5244 or toll free at 1-866-680-2906. You can also write to the Stanford IRB, Stanford University, 1705 El Camino Real, Palo Alto, CA 94306.

#### **FUTURE PARTICIPATION**

The researchers may want to contact you after your participation in this project ends. They may want to get more information or perform more procedures for this project or they may want to ask you and/or your child to participate in another project. You should indicate below whether or not you agree to allow the study staff to contact you for these reasons by placing an "X" by the appropriate statement. Your answer will not affect your ability or anyone else's to participate in this study. If you change your mind at any time, please contact the study staff.

| I agree to allow the study staff to contact me if they need more information from me for this study or if they would like to offer me participation in another project. |
|---|
| I do not want the study staff to contact me after I finish participating in this study. |

IRB Use Only

Approval Date: November 30, 2022 Expiration Date: November 30, 2023

Protocol Director: Kimford Meador, MD

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

**EXPERIMENTAL SUBJECTS BILL OF RIGHTS:** As a research participant you have the following rights. These rights include but are not limited to the participant's right to:

- be informed of the nature and purpose of the experiment;
- be given an explanation of the procedures to be followed in the medical experiment, and any drug or device to be utilized;
- be given a description of any attendant discomforts and risks reasonably to be expected;
- be given an explanation of any benefits to the subject reasonably to be expected, if applicable;
- be given a disclosure of any appropriate alternatives, drugs or devices that might be advantageous to the subject, their relative risks and benefits;
- be informed of the avenues of medical treatment, if any available to the subject after the experiment if complications should arise;
- be given an opportunity to ask questions concerning the experiment or the procedures involved;
- be instructed that consent to participate in the medical experiment may be withdrawn at any time and the subject may discontinue participation without prejudice;
- be given a copy of the signed and dated consent form; and

The extra copy of this signed and dated consent form is for you to keep.

• be given the opportunity to decide to consent or not to consent to a medical experiment without the intervention of any element of force, fraud, deceit, duress, coercion or undue influence on the subject's decision.

| ,, , | , . |
|---|---|
| Signature of Adult Participant | <br>Date |
| Print Name of Adult Participant | |
| Signature of Legally Authorized Representative (LAR) (e.g., parent, guardian or conservator) | Date |
| Print Name of LAR | |
| LAR's Authority to Act for Participant (e.g. parent guardian or conservator) | |

IRB Use Only

Approval Date: November 30, 2022 Expiration Date: November 30, 2023

Protocol Director: Kimford Meador, MD

Protocol Title: Maternal Outcomes and Neurodevelopmental Effects of Antiepileptic Drugs (MONEAD) V7.2-Mother

| (If available) Signature of Other Parent or Gua | ardian Date |
|---|---|
| Print Name of Other Parent or Guardian | |
| Authority to Act for Participant | |
| Signature of Person Obtaining Consent | Date |
| Print Name of Person Obtaining Consent | |
| The following witness line is to be signed only if the accompanied by a short form foreign language co | · |
| Signature of Witness | <br>Date |
| Print Name of Witness | |

(e.g., staff, translator/interpreter, family member, or other person who speaks both English and the participant's language)

- Translated short form must be signed and dated by both the participant (or their LAR) AND the witness.
- The English consent form (referred to as the "Summary Form" in the regulations):
  - o Must be signed by the witness AND the Person Obtaining Consent (POC).
  - o The non-English speaking participant/LAR does not sign the English consent.
  - o The non-English speaking participant/LAR should not sign the HIPAA participant line
  - If the participant or the LAR is non-English speaking, the Person Obtaining Consent (POC) must ensure that 1) the LAR's Description of Authority is completed and 2) that any questions or options presented by the consent form are documented and initialed by the POC on the Summary Form, per the participant's wishes, as they are understood during the consent process.